CLINICAL TRIAL: NCT03146442
Title: Increased Protein at Breakfast for Weight Management in Overweight Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: University of Kansas Medical Center (Other); University of Tennessee (Other)
Responsible Party: Principal Investigator, Heather Leidy, Associate Professor, University of Texas at Austin
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: 1611018490
Record Dates: First submitted 2017-05-07; First posted 2017-05-10 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Obesity, Adolescent
Keywords: increased dietary protein; breakfast; weight management; satiety; glucose control; fMRI; cognitive performance; memory; attention; executive function; structural MRI; sleep quality
MeSH Terms: conditions — Pediatric Obesity; Sleep Initiation and Maintenance Disorders | interventions — Breakfast

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to the following breakfast groups: high protein breakfast (350kcal; 34% protein (30g protein), 40% CHO, and 26% fat); normal protein breakfast (350kcal; 11% protein (10g protein), 63% CHO, and 26% fat); or breakfast skipping (0 kcal)
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blind, the PI and outcomes assessor will be blinded to the intervention arms (which will be designated with code words). The participants in the high protein and normal protein intervention arms will be blinded to the protein content within the breakfast meals (which will be designated with code words).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Normal Protein (NP) Breakfast (Active Comparator): The participants in the NP Breakfast group will be provided with NP Breakfasts to consume, at home, between 6:00-9:00 am each day over the 6-month intervention. The energy content of the breakfast meals will be standardized to 350 kcal. The energy content of the breakfast meals is ~18% of daily energy intake estimated from the energy expenditure equations specific for adolescents ages 13-19y. The NP breakfasts will be 11% protein (10g protein), 63% CHO, and 26% fat. The types of protein incorporated within the NP and HP meals will include a combination of animal (egg, dairy, animal tissue) and plant-based proteins (soy, pea, gluten). An 8-d breakfast rotation will occur throughout the 6 months.
  Interventions: Behavioral: Breakfast
- High Protein (HP) Breakfast (Experimental): The participants in the HP Breakfast group will be provided with HP Breakfasts to consume, at home, between 6:00-9:00 am each day over the 6-month intervention. The energy content of the breakfast meals will be standardized to 350 kcal. The energy content of the breakfast meals is ~18% of daily energy intake estimated from the energy expenditure equations specific for adolescents ages 13-19y. The HP breakfasts will be 34% protein (30g protein), 40% CHO, and 26% fat. The types of protein incorporated within the HP and HP meals will include a combination of animal (egg, dairy, animal tissue) and plant-based proteins (soy, pea, gluten). An 8-d breakfast rotation will occur throughout the 6 months.
  Interventions: Behavioral: Breakfast
- Breakfast Skipping (BS) (Placebo Comparator): The participants in the BS group will continue to skip breakfast each day over the 6-month intervention. They will have nothing to eat or drink (besides water) until 11 am.
  Interventions: Behavioral: Breakfast

INTERVENTIONS:
Behavioral: Breakfast — For 6 months, the participants will either skip breakfast or will habitually consume a NP or HP breakfast every day.

SUMMARY:
Adolescent obesity, negatively affecting the lives of over 18 million (34%) US adolescents, continues to be a major public health concern due to the increased risk of developing chronic diseases, including type 2 diabetes. Thus, there is a great need to develop effective, dietary strategies that target health outcomes, including weight management and glycemic control in young people. One particular strategy that is gaining scientific support includes the daily consumption of a protein-rich breakfast. This study will identify the potential role of protein at breakfast as a key component of a healthy diet for improvements in appetite control, satiety, and weight management to reverse the obesity epidemic and prevent and/or delay serious health complications in young people.

DETAILED DESCRIPTION:
Adolescent obesity continues to be a major public health concern due to the increased risk of developing chronic diseases, including, but not limited to, type 2 diabetes. Thus, strategies are vitally needed that target weight management and glycemic control to reverse the obesity epidemic and prevent and/or delay serious health complications in young people. The daily consumption of breakfast has been touted as an essential part of the diet to prevent and/or treat obesity. While breakfast was once thought to be 'the most important meal of the day', this notion has recently been challenged due to the paucity of existing causal evidence. In addition, interest in the study of breakfast and weight management has highlighted the importance of macronutrient content, particularly increased dietary protein at breakfast, as a critical factor. Pilot data has illustrated reductions in body fat mass and improvements in glycemic control following the daily consumption of high protein breakfasts over a short period in overweight adolescents. However, it is unclear as to whether these effects would occur over the long-term and what mechanisms-of-action contribute to the improvements in these health outcomes. Aim 1 will determine whether a causal link exists between breakfast, particularly one rich in dietary protein, and weight management in young people. To accomplish this, 150 overweight, habitual breakfast-skipping adolescents will complete the following long-term randomized, tightly-controlled breakfast trial. Participants will be randomly provided with high protein breakfasts (350kcal; 34% protein (30g protein), 40% CHO, and 26% fat); isocaloric normal protein breakfasts (350kcal; 11% protein (10g protein), 63% CHO, and 26% fat); or will continue to skip breakfast for 6 mo. Baseline, 3, and 6 body weight, body composition, and free-living glycemic control will be assessed. In addition, daily intake, with particular focus on evening snacking behavior, will also be measured at baseline, 3, and 6 mo. Aim 2 will identify the appetitive, hormonal, and neural signals by which a protein breakfast modulates ingestive (i.e., eating) behavior and weight management. To address this aim, a sub-set of the 150 (n=75) will complete 10-h testing days during baseline, 3, and 6 mo. Repeated assessments of perceived appetite, satiety, and food cravings along with appetite-regulating hormonal responses (i.e., plasma ghrelin, GLP-1, PYY, and HVA (the primary dopamine metabolite)) will be measured throughout the day. In addition, post-breakfast and pre-dinner functional (fMRI) brain scans will also be completed to identify neural activation to food stimuli in cortico-limbic brain regions known to modulate food motivation, reward, and cravings along with structural scans. Aim 3 will identify specific appetitive, hormonal, and neural signals as strong predictors of ingestive behavior and weight management. Within this sub-set of 150, aim 4 will determine whether a causal link exists between breakfast, particularly one rich in dietary protein, and cognitive performance (memory, attention, and executive function). These assessments will also be paired with structural scans. The measures collected in Aim 2 will be analyzed in combination with food choice, daily intake, weight loss, and reductions in body fat following the 6-mo interventions. Collectively, this project will provide novel evidence testing the consumption of a high protein breakfast as a dietary strategy to combat obesity in young people.

ELIGIBILITY:
Inclusion Criteria:

* All ethnicities
* BMI: 25-34kg/m2 or 85th-98th percentile
* Skips Breakfast (<110 kcal prior to 10 am) at least 4 days/week for the past year
* Never smoked or used other tobacco products
* Willing to consume the study breakfasts
* Generally healthy

Exclusion Criteria:

* Clinically diagnosed with an eating disorder
* Metabolic, hormonal, and/or neural conditions/diseases that influence metabolism or appetite
* Currently or previously on a weight loss or other special diet (in the past 6 months)
* Gained/lost ≥4.5kg over the past 6 months
* Taking medication that would directly influence appetite (weight-loss drugs or antidepressant, steroid, or thyroid medication, unless dosage has been stable for at least 6 months)
* Normal cognitive restraint (assessed from the Three Factor Eating Habits Questionnaire)
* Does not consistently eat lunch and/or dinner every day

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 103 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Fat Mass Change | Baseline, 3 month, and 6 month
  Whole body fat mass will be determined with Dual X-ray Absorptiometry (DXA). The DXA uses a linear X-ray fan beam with switched-pulse dual-energy and a multi-element detector array. The whole body scan takes <1.8 sec with radiation exposure of 0.01mGy.
3-day Average Daily Intake Change | Baseline, 3 month, and 6 month
  Free-living daily energy intake will be assessed for 3 consecutive days through daily food packouts. The participants will be provided with an excess of macronutrient-specific meals, snacks, and beverages to consume, ad libitum, throughout each day in addition to the required, respective breakfast treatment. The quantity of food provided will be ~50% more than their estimated, weight-maintaining energy intake. All food items will be initially weighed and recorded. The participants will be instructed to return all uneaten foods as well as all wrappers and containers from consumed food. Any partially eaten, returned items will be weighed accordingly. Daily energy content will be assessed from these packouts.
Glucose Excursions Change | Baseline, 3 month, and 6 month
  Free-living, glucose measures will be performed for 6 consecutive days using Continuous Glucose Monitoring Device. The participants will report to our facility during one afternoon for insertion. A small area on the participant's abdomen will be cleaned and the tiny glucose sensor will be inserted just under the skin and held in place with Tegederm. The sensor measures glucose every 10sec and records an average glucose value every 5min for up to 144h.Calibration is performed by 4 finger sticks/d with a glucose analyzer.
PYY Change | Baseline, 3 month, and 6 month
  During a single clinical visit, 22 blood samples (4 ml/sample) will be collected throughout a 10-h period. The samples will be collected in EDTA test tubes containing pefabloc SC and DPP-IV to reduce protein degradation. Within 10-min of collection, the samples will be centrifuged, and the plasma will be stored at -80°C for future analysis. Plasma total PYY will be measured using magnetic bead-based multi-analyte assays (Millipore, St.Charles, MO) & Luminex technologies (Luminex Corporation, Austin, TX).
Fullness Change | Baseline, 3 month, and 6 month
  During a single clinical visit, 22 questionnaires, assessing feelings of 'fullness' will be collected over a 10-h period. The questionnaires contain VAS incorporating a 100mm horizontal line rating scale for each response. The questions are worded as "how strong is your feeling of" with anchors of "not all" to "extremely." The Adaptive Visual Analog Scale Software will be used for data collection (Neurobehavioral Research Laboratory and Clinic; San Antonio, TX).
Cravings for Fats Change | Baseline, 3 month, and 6 month
  During a single clinical visit, 22 questionnaires, assessing cravings for fat foods will be collected over a 10-h period. The questionnaires contain VAS incorporating a 100mm horizontal line rating scale for each response. The questions are worded as "how strong is your feeling of" with anchors of "not all" to "extremely." The Adaptive Visual Analog Scale Software will be used for data collection (Neurobehavioral Research Laboratory and Clinic; San Antonio, TX).
fMRI Anterior Cingulate Neural Response Change | Baseline, 3 month, and 6 month
  During a single clinical visit, the participants will arrive at the testing facilities 1-h prior to breakfast, following a 10-h overnight fast. The participants will be taken to a self-contained, comfortable, quiet room. At +0 min, the participants will consume the respective breakfast (or continue to skip breakfast). Immediately after breakfast, the participants will complete a food cue-stimulated fMRI brain scan. After the completion of the scan participants will complete the remaining testing procedures. At approximately 4-h after breakfast the participants will be provided with a standardized lunch and then continue with testing procedures. 3.5-h following lunch, participants will complete a final fMRI brain scan.

SECONDARY OUTCOMES:
Sleep Health | Baseline, 3 month, and 6 month
  Free-living sleep will be measured for 7 days through actigraphy. The device will be worn on the wrist for 7 days and the participant will continuously wear it over the next 7 days for an overall measurement of sleep quality. Sleep quality and daytime sleepiness will also be assessed using sleep diaries and questionnaires.
Cognitive Function | Baseline, 3 month, and 6 month
  During a single clinical visit, the participants will arrive at the testing facilities 1-h prior to breakfast, following a 10-h overnight fast. The participants will be taken to a self-contained, comfortable, quiet room. 30 minutes prior to breakfast, participants will begin a series of cognitive tests assessing memory, attention, and executive function. At +0 min, the participants will consume the respective breakfast (or continue to skip breakfast). At +90 and +150 min, participants will complete the same series of cognitive tests assessing memory, attention, and executive function.
Structural MRI Change | Baseline and 6 month
  During a single clinical visit, the participants will arrive at the testing facilities 1-h prior to breakfast, following a 10-h overnight fast. The participants will be taken to a self-contained, comfortable, quiet room. At +0 min, the participants will consume the respective breakfast (or continue to skip breakfast). After breakfast, the participants will complete a brain scan that includes structural analysis.
Cortisol Change | Baseline, 3 month, and 6 month
  Salivary samples will be collected prior to sleep onset and upon waking at various times throughout baseline, 3-month, and 6-month testing periods. The samples will be collected in mini cryo-tubes and stored at -80°C for future analysis. Salivary cortisol will be measured using a competitive immunoassay designed and validated for the quantitative determination of melatonin in saliva (Salimetrics, State College, PA).
Melatonin Change | Baseline, 3 month, and 6 month
  Salivary samples will be collected prior to sleep onset and upon waking at various times throughout baseline, 3-month, and 6-month testing periods. The samples will be collected in mini cryo-tubes and stored at -80°C for future analysis. Salivary melatonin will be measured using a competitive immunoassay designed and validated for the quantitative determination of melatonin in saliva (Salimetrics, State College, PA).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Piacquadio KA, Margolis LM, Gwin JA, Leidy HJ. Preliminary Evidence Supports that Long-Term Consumption of Higher-Protein Breakfast Promotes Higher Expression of Select miRNA Associated with Cardiometabolic Health in Adolescents. J Nutr. 2024 Dec;154(12):3585-3591. doi: 10.1016/j.tjnut.2024.10.007. Epub 2024 Oct 10. PMID 39393494